CLINICAL TRIAL: NCT06639555
Title: Initial Clinical and CBCT Outcomes of Enamel Matrix Derivative-Based Regenerative Therapy in Vertical Bone Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsvetalina Gerova-Vatsova (Other)
Responsible Party: Sponsor-Investigator, Tsvetalina Gerova-Vatsova, Assistant, Medical University of Varna
Organization: Medical University of Varna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118/23.06.22
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vertical Alveolar Bone Loss
MeSH Terms: interventions — emerin; Guided Tissue Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PRP alone (Active Comparator)
  Interventions: Procedure: PRP( platelet rich plasma)
- EMD Alone (Active Comparator)
  Interventions: Procedure: EMD (Enamel Matrix Derivative)
- GTR (barrier membrane) (Active Comparator)
  Interventions: Procedure: Guided Tissue Regeneration (barrier membrane)
- GTR(barrier membrane and PRP) (Active Comparator)
  Interventions: Procedure: Guided Tissue Regeneration(barrier membrane and PRP)

INTERVENTIONS:
Procedure: PRP( platelet rich plasma) — regenerative therapy with PRP for vertical bone defects
  Arms: PRP alone
Procedure: EMD (Enamel Matrix Derivative) — regenerative therapy with EMD for vertical bone defects
  Arms: EMD Alone
Procedure: Guided Tissue Regeneration (barrier membrane) — guided tissue regeneration with barrier membrane alone for vertical bone defects
  Arms: GTR (barrier membrane)
Procedure: Guided Tissue Regeneration(barrier membrane and PRP) — guided tissue regeneration with barrier membrane and PRP for vertical bone defects
  Arms: GTR(barrier membrane and PRP)

SUMMARY:
Study of the effectiveness of the application of regenerative therapy with autogenous, platelet-rich plasma in vertical defects Investigation of the effectiveness of the application of regenerative therapy with enamel matrix derivatives in vertical bone defects Study of the effectiveness of the application of guided tissue regeneration in vertical bone defects with Barrier membrane and Barrier membrane and autogenous platelet-rich plasma

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* written informed consent
* age
* no systemic diseases

Exclusion Criteria:

* smokers
* horizontal bone loss
* untreated periodontium disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Probing depth in mm | 6 months
Level of Margo Gingivalis in mm | 6 months
Clinical attachment level in mm | 6 months
The distance from the ECJ to the base of the bone defect in mm | 6 months
The distance from the ECJ to the apex of the bone defect in mm | 6 months
The width of the bone defect in mm | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University - Varna, Varna, Varna, Bulgaria